CLINICAL TRIAL: NCT04864054
Title: An Open-Label, Dose Escalation, Multi-Center Phase I/II Clinical Trial of ECT204 T-Cell Therapy in Adults With Advanced Hepatocellular Carcinoma (HCC) (ARYA-3)
Brief Title: T-Cell Therapy (ECT204) in Adults With Advanced HCC
Acronym: ARYA-3
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eureka Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETUS20GPC3AR124
Record Dates: First submitted 2021-04-14; First posted 2021-04-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer, Adult; Liver Neoplasm; Metastatic Liver Cancer
Keywords: Hepatocellular Carcinoma; Advanced HCC; Late-Stage HCC; Liver Cancer; Liver Neoplasm; Metastatic Liver Cancer; Metastatic HCC; T-cell therapy; Immunotherapy; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation, RP2D Confirmatory, and Expansion (Phase 1/2 Single Arm) (Experimental): Dose Escalation Cohort: Patients receive a single infusion of ECT204 T cells at one of four predefined dose levels on Day 0 after conditioning. Conditioning consists of fludarabine (Flu) and cyclophosphamide (Cy).
  RP2D Confirmatory Cohort: Patients receive ECT204 T cells at the RP2D on Day 0 and may receive a second infusion approximately one month later. This cohort uses the same Flu/Cy conditioning as the dose-escalation cohort; no conditioning is given before the second ECT204 infusion.
  Expansion Cohort: Patients receive multiple ECT204 infusions at the RP2D (initial on Day 0, planned second on Day 31, and optional third or later doses). The third infusion may be administered no earlier than Day 60, and each subsequent infusion must be separated by at least 30 days. Patients receive Flu/Cy/regorafenib before the first infusion and regorafenib alone before the second and subsequent infusions.
  Interventions: Biological: ECT204 T cells

INTERVENTIONS:
Biological: ECT204 T cells — ECT204 is an autologous T-cell therapy whereby a subject's own T cells are transduced with a lentiviral vector expressing the ECT204 transgene.

SUMMARY:
This is an open-label, dose escalation, multi-center, Phase I/II clinical trial aimed at assessing the safety and preliminary efficacy of an investigational ARTEMIS® ECT204 T-cell therapy. The trial is suitable for adult subjects (≥ 18 years of age) diagnosed with GPC3-positive HCC, who have failed or not tolerated at least two (2) different anti-HCC systemic agents.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation, multi-center, Phase I/II clinical trial. The purpose of this study is to evaluate an investigational ECT204 T-cell therapy in adult patients with GPC3-positive advanced hepatocellular carcinoma (HCC). ECT204 is an autologous T-cell product built on the ARTEMIS® cell receptor platform that involves two GPC3-targeting surface components: an antibody-T-cell receptor (AbTCR) and a chimeric stimulating receptor (CSR; also referred to as the co-stimulatory molecule). In this study, T cells are collected from each patient and genetically modified ex vivo to co-express the GPC3-specific AbTCR and GPC3-specific CSR, then re-administered to the patient to selectively recognize and eliminate GPC3-expressing HCC tumor cells.

The protocol describes two parts: Part 1 (dose escalation) and Part 2 (expansion).

Part 1: Dose Escalation

Part 2: Expansion

- The initial cohort of Part 2 is defined as the "RP2D Confirmatory Cohort"

'Phase 1' is defined as Part 1 plus the initial RP2D confirmatory cohort in Part 2, and 'Phase 2' is defined as the subsequent expansion cohort in Part 2.

The protocol itself does not label phases; it uses Part 1 and Part 2 terminology only.

The active assessment period of the study will continue for 2 years. Subjects will be followed for assessment of treatment safety and overall survival during Long Term Follow-Up (LTFU; year 2 -15).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HCC, that is unresectable, recurrent, and/or metastatic.
* GPC3-positive tumor expression confirmed by immunohistochemistry (IHC).

  * For the dose-escalation cohort: ≥10-20% tumor cells, ≥2+ IHC.
  * Beginning with the RP2D confirmatory cohort: ≥ 50% tumor cells, 2+/3+ IHC.
* Must have failed, or not tolerated, at least two (2) different anti-HCC systemic agents.
* Life expectancy of at least 4 months per the Investigator's opinion.
* Karnofsky Performance Scale of 70 or higher.
* Measurable disease by RECIST v1.1.
* Child-Pugh score of A6 or better.
* Adequate organ function.

Exclusion Criteria:

* Pre-existing illness (e.g., symptomatic congestive heart failure) that would limit compliance with study requirements.
* Active, uncontrolled systemic bacterial, fungal, or viral infection. Subjects with Human Immunodeficiency Virus (HIV), hepatitis B, or hepatitis C are eligible provided their infection is being treated and the viral load is controlled.
* Active malignancy (other than HCC), with the exception of cholangiocarcinoma (CCA) or any malignancy without any organ involvement and with an expected survival ≥ 3 years without any treatment (exception: hormone/androgen- deprivation therapy).
* Pregnant or lactating women.
* Currently receiving or ending (< 14 days from date of consent) liver tumor-directed therapy (e.g., radiation, ablation, embolization), or hepatic surgery.
* Concurrently receiving other investigational agents, biological, chemical, or radiation therapies, while participating in the study.
* Active autoimmune disease requiring systemic immunosuppressive therapy.
* Presence of portal vein tumor thrombus (PVTT) classified as grade Vp4, or any invasion into the inferior vena cava (IVC).
* Ascites requiring active treatment.
* History of organ transplant.
* Advanced HCC involving greater than half (50%) of the liver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and tolerability of ECT204 in adult subjects with advanced HCC | Up to 2 years (active assessment period); additional long-term follow-up (LTFU) up to 15 years
  Type, frequency, and severity of adverse events (AEs) and laboratory abnormalities
Determine the Recommended Phase II Dose (RP2D) of ECT204 (Concluded During Phase 1 of the study) | Up to 28 days
  RP2D determination is based on the maximum tolerated dose (MTD), defined as the highest dose level at which the proportion of subjects experiencing a Dose-Limiting Toxicity (DLT) is less than or equal to 30% and does not exceed the maximum administered dose (MAD). Final determination is based on the observed DLT rates and manufacturing capability, and is made by the Dose Escalation Committee (DEC).

SECONDARY OUTCOMES:
Assess the efficacy of ECT204 in adult subjects with advanced HCC using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (RECIST v1.1) as the primary criterion. | Up to 2 years
  Overall Response Rate (ORR), defined as the proportion of subjects with a best overall response (BOR) of either complete response (CR) or partial response (PR).
Assess the efficacy of ECT204 | Disease Control Rate | Up to 2 years
  Disease Control Rate (DCR), defined as the proportion of subjects with BOR of either CR, PR, or stable disease (SD).
Assess the efficacy of ECT204 | Duration of Response | Up to 15 years
  Duration of Response (DOR), defined as the time from first response to progressive disease (PD) or death.
Assess the efficacy of ECT204 | Progression-Free Survival | Up to 15 years
  Progression-Free Survival (PFS), defined as the time from ECT204 infusion to PD or death
Assess the efficacy of ECT204 | Time to Progression (TTP) | Up to 15 years
  Time to Progression (TPP), defined as the time from ECT204 infusion to the date of death.
Assess the efficacy of ECT204 | Overall Survival | Up to 15 years
  Overall Survival (OS), defined as the time from ECT204 T-cell infusion to the date of death.
Characterize the pharmacokinetic (PK) profile of ECT204, including the expansion and persistence of ECT204, in our study subject population | Peak Exposure (Cmax) | Up to 2 years
  The peak exposure (Cmax) will be measured.
Characterize the pharmacokinetic (PK) profile of ECT204, including the expansion and persistence of ECT204, in our study subject population | Time to reach peak exposure (Tmax) | Up to 2 years
  The time to reach peak exposure (Tmax) will be measured.
Characterize the pharmacokinetic (PK) profile of ECT204, including the expansion and persistence of ECT204, in our study subject population | Partial area under the curve (pAUC) | Up to 2 years
  The partial area under the curve (pAUC) will be measured.
Characterize the pharmacokinetic (PK) profile of ECT204, including the expansion and persistence of ECT204, in our study subject population | Other relevant PK parameters in peripheral blood (PB) | Up to 2 years
  Other relevant PK parameters of ECT204 in peripheral blood (PB) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Pei Wang, PhD, Study Director — Eureka Therapeutics Inc.
Locations (7):
- United States (6):
  - City of Hope, Duarte, California
  - Kansas University Medical Center, Principal Investigator:, Westwood, Kansas
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Texas Southwestern, Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - Fred Hutchinson Cancer Center, University of Washington, Seattle, Washington
- National Taiwan University Cancer Center, Taipei, Taiwan